CLINICAL TRIAL: NCT05986630
Title: A Prospective, Randomized, Blinded Evaluator, Multicenter, Clinical Study to Evaluate Safety and Effectiveness of TEOSYAL® TPVM Versus COMPARATOR for the Remodeling of the Lower Face
Brief Title: Safety and Effectiveness Evaluation of TEOSYAL® TPVM Versus COMPARATOR for the Remodeling of the Lower Face
Acronym: LIFTUP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEO-TPVM-2101
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Aging; Chin Retrusion
Keywords: Dermal filler; Hyaluronic acid (HA); Chin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEOSYAL® TPVM (Experimental): n=116 subjects
  Interventions: Device: TEOSYAL® TPVM
- COMPARATOR (Active Comparator): n= 39 subjects
  Interventions: Device: COMPARATOR

INTERVENTIONS:
Device: TEOSYAL® TPVM — Injection of TEOSYAL® TPVM at Baseline
  Optional Touch-up treatment at 4 weeks if needed to achieve optimal correction as judged by the PI.
  Arms: TEOSYAL® TPVM
Device: COMPARATOR — Injection of a COMPARATOR at Baseline
  Optional Touch-up treatment at 4 weeks if needed to achieve optimal correction as judged by the PI.
  Arms: COMPARATOR

SUMMARY:
The clinical study is designed to prospectively evaluate the safety and effectiveness of TEOSYAL® TPVM when compared to COMPARATOR for the remodeling of the lower face

DETAILED DESCRIPTION:
This is a prospective, randomized, blinded evaluator, multicenter, clinical study to evaluate safety and effectiveness of TEOSYAL® TPVM versus COMPARATOR for the remodeling of the lower face.

Subject will be enrolled in the study based on evaluation of their chin retrusion severity.

For the purpose of this study, all injections will be done by principal investigators (PIs) with several years of experience in aesthetic treatment.

An external aesthetic and cosmetic surgeon will act as a BE to assess the performance of the treatment and the product based on photographs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects over 18 years old seeking correction of their lower face
* Subject scored grade 2 or 3 on the TCRS
* Female subjects of childbearing potential must have a negative UPT and practice a reliable method of contraception throughout the study.
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations
* Able to follow study instructions and complete all required visits.
* Having given its signed informed consent

Exclusion Criteria:

* Known hypersensitivity or previous allergic reaction to any component of the study devices
* Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
* History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
* Subject exhibits any physical attribute that may prevent assessment or treatment of the lower face as judged by the PI
* Clinically significant alcohol or drug abuse.
* Subject has received any investigational product within 90 days prior to Visit 1 or planning to participate in another investigation during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in TCRS score between Baseline and 8 weeks after last treatment as assessed by the Blinded Evaluator | 8 weeks
  Non-inferiority of TCRS score change from Baseline for subjects treated with TEOSYAL TPVM compared to subjects treated with a COMPARATOR at 8 weeks after last treatment as assessed by the BE.
  TCRS (Teoxane Chin Retrusion Scale) is a validated 4-point scale assessing chin retrusion severity with 0 being "None/minimal" and 3 being "Severe"

CONTACTS AND LOCATIONS:
Locations (1):
- Care- Geneva, Geneva, Switzerland